CLINICAL TRIAL: NCT04653675
Title: Cardiac Amyloidosis in Spinal Stenosis: the CASS-study
Acronym: CASS
Status: Active, not recruiting | Type: Observational
Sponsor: AZ Sint-Jan AV (Other)
Responsible Party: Principal Investigator, Philippe Debonnaire, Principal Investigator, AZ Sint-Jan AV
Other Study IDs: 2741
Record Dates: First submitted 2020-11-19; First posted 2020-12-04 (Actual); Last update posted 2024-08-07 (Actual); Status verified 2024-08

CONDITIONS: Cardiac Amyloidosis
MeSH Terms: conditions — Amyloid Neuropathies, Familial

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Background: A significant portion of cardiac amyloidosis patients have a 5 to 10 years prior history of spinal canal stenosis, reflecting a diagnostic red flag that should raise suspicion for amyloidosis presence. Mild troponin release and NT-proBNP elevation, both serum cardiac biomarkers, often coincide with cardiac amyloidosis. Early cardiac amyloidosis treatment improves survival, warranting timely diagnosis.

Study aim: to test a prospective screening strategy, based on serum cardiac biomarkers, to increase early detection of cardiac amyloidosis in patients with spinal canal stenosis.

Design: Single-centre prospective observational non-interventional diagnostic study.

Methods: Consecutive patients during a one-year period in AZ Sint-Jan Bruges, without known cardiac amyloidosis history and scheduled for spinal canal stenosis surgery, will have cardiac evaluation including serum cardiac biomarker (high-sensitive troponin T and NT-proBNP) assessment, electrocardiography and transthoracic echocardiography. During surgery, all patients will undergo ligamentum flavum biopsy to evaluate presence and burden of transthyretin amyloid deposition (Congo-red staining and immune histochemistry). All patients with suspicion for cardiac amyloidosis will undergo further diagnostic testing (including laboratory test and bone scintigraphy). A chronologic cascade screening process will be used starting with abnormal serum cardiac biomarkers (high-sensitive troponin T ≥ 14 ng/ml and/or NT-proBNP > 125 pg/ml), followed by electrocardiography, transthoracic echocardiography and finally ligamentum flavum biopsy results. The diagnostic performance of this biomarker-based strategy will be compared to electrocardiography, echocardiography and ligamentum flavum biopsy.

Conclusion: It is hypothesised that serum cardiac biomarker testing in patients undergoing spinal canal stenosis surgery represents a simple and valuable prospective screening strategy for early detection of cardiac amyloid(osis).

ELIGIBILITY:
Inclusion Criteria:

* Cervical or lumbar spinal canal stenosis, scheduled for spinal surgery
* > 18 years old

Exclusion Criteria:

Prior diagnosis of cardiac amyloidosis and evident alternative explanations for troponin and/or NT-proBNP elevation are the main reasons for exclusion.

* known cardiac amyloidosis
* severe valvular regurgitation or stenosis
* Left ventricular ejection fraction (LVEF) < 40%
* Glomerular filtration rate (GFR) ≤ 25 ml/kg/min or dialysis
* recent heart failure admission ≤ 1 month
* recent myocarditis ≤ 3 months
* recent acute coronary syndrome ≤ 1 month
* recent percutaneous coronary intervention (PCI) ≤ 1 month
* recent cardiac surgery ≤ 3 months
* active or planned pregnancy
* unwilling to participate or provide signed informed consent

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with cervical or lumbar spinal canal stenosis scheduled for spinal surgery
Sampling Method: Probability Sample
Enrollment: 105 (Actual)
Dates: Start 2021-01-01 (Actual); Primary Completion 2022-06-30 (Actual); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
Diagnostic performance hs-Troponin T (ng/L) to early diagnose cardiac amyloidosis | 12 months after spinal canal surgery
  Diagnostic performance of a prospective screening strategy, based on elevated hs-Troponin T (ng/L), in patients with spinal canal stenosis undergoing spinal surgery, to early diagnose cardiac amyloidosis
Diagnostic performance of NT-proBNP (pg/ml) to early diagnose cardiac amyloidosis | 12 months after spinal canal surgery
  Diagnostic performance of a prospective screening strategy, based on elevated NT-proBNP (pg/ml), in patients with spinal canal stenosis undergoing spinal surgery, to early diagnose cardiac amyloidosis
Difference in diagnostic performance of NT-proBNP (pg/ml) and echocardiography, electrocardiography and ligamentum flavum biopsy | 12 months after spinal canal surgery
  Difference in diagnostic performance of NT-proBNP (pg/ml) with CA suspicion based on echocardiography (left ventricular wall thickness), electrocardiography (QRS amplitude, presence of atrial fibrillation) and ligamentum flavum biopsy (presence of transthyretin-amyloid deposits)

SECONDARY OUTCOMES:
Difference in diagnostic performance of hs-Troponin T (ng/L) and electrocardiography parameters | 12 months after spinal canal surgery
  Difference in diagnostic performance of hs-Troponin T (ng/L) with CA suspicion based on electrocardiography (QRS amplitude, presence of atrial fibrillation)
Difference in diagnostic performance of hs-Troponin T (ng/L) and echocardiography parameters | 12 months after spinal canal surgery
  Difference in diagnostic performance of hs-Troponin T (ng/L) with CA suspicion based on echocardiography (left ventricular wall thickness)
Difference in diagnostic performance of hs-Troponin T (ng/L) and ligamentum flavum biopsy | 12 months after spinal canal surgery
  Difference in diagnostic performance of hs-Troponin T (ng/L) with CA suspicion based on ligamentum flavum biopsy (presence of transthyretin-amyloid deposits)
Difference in diagnostic performance of NT-proBNP (pg/ml) and echocardiography parameters | 12 months after spinal canal surgery
  Difference in diagnostic performance of NT-proBNP (pg/ml) with CA suspicion based on echocardiography (left ventricular wall thickness)
Difference in diagnostic performance of NT-proBNP (pg/ml) and electrocardiography parameters | 12 months after spinal canal surgery
  Difference in diagnostic performance of NT-proBNP (pg/ml) with CA suspicion based on electrocardiography (QRS amplitude, presence of atrial fibrillation)
Difference in diagnostic performance of NT-proBNP (pg/ml) and ligamentum flavum biopsy | 12 months after spinal canal surgery
  Difference in diagnostic performance of NT-proBNP (pg/ml) with CA suspicion based on ligamentum flavum biopsy (presence of transthyretin-amyloid deposits)
To determine the prevalence of TTR amyloid in both cervical and lumbar spinal canal stenosis patients as function of age and clinical presentation | 6 months after spinal canal surgery
To correlate TTR amyloid burden on ligamentum flavum biopsy to echocardiographic (e.g. ventricular wall thickness) parameters | 12 months after spinal canal surgery
To correlate TTR amyloid burden on ligamentum flavum biopsy to cardiac biomarker parameters (e.g. hs-Troponin T (ng/L)) | 12 months after spinal canal surgery

CONTACTS AND LOCATIONS:
Overall Officials: Philippe Debonnaire, MD, PhD, Principal Investigator — AZ Sint-Jan AV
Locations (1):
- AZ Sint-Jan Brugge-Oostende AV, Bruges, Belgium